CLINICAL TRIAL: NCT02919332
Title: Improved Visualization of Glioblastoma Using Delayed 18F-FDG PET/CT.
Brief Title: Delayed 18F-FDG PET/CT in Improving Visualization of Brain Tumors in Patients With Glioblastoma
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-000600; NCI-2016-01214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID655 (Other: UCLA / Jonsson Comprehensive Cancer Center); 16-000600 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2016-08-30; First posted 2016-09-29 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma; Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic (18F-FDG PET/CT): Patients receive fludeoxyglucose F-18 IV. Patients then undergo a standard of care PET/CT scan at 60 minutes and a second PET/CT scan at 240 minutes after injection.
  Interventions: Procedure: Computed Tomography; Radiation: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 18F-FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Radiation: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo 18F-FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies how well delayed fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET)/computed tomography (CT) works in improving visualization of brain tumors in patients with glioblastoma. Radiotracers such as 18F-FDG are highly taken up by tumors in the brain and are visualized using PET/CT. Increasing the interval of time between 18F-FDG administration and PET/CT scan may improve the visualization of brain tumors in patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve the visualization/delineation of glioblastoma lesions using delayed 18F-FDG PET/CT imaging.

OUTLINE:

Patients receive fludeoxyglucose F-18 intravenously (IV). Patients then undergo a standard of care PET/CT scan at 60 minutes and a second PET/CT scan at 240 minutes after injection.

Note:

Standard Uptake Value (SUV) is defined for state-of-the art PET/CT scanners as Standardized uptake values = count activity per ml within region of interest (MBq/ml)/[injected dose (MBq)/body weight (kgx1000)]

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven high grade glioma scheduled for 18F-FDG PET/CT

Exclusion Criteria:

* Severe psychiatric illness
* Inability to give written consent
* Breast feeding/pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age who have been diagnosed with a brain tumor and are undergoing a PET/CT scan..
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Tumor-to-background ratio on delayed scans (240 min after injection) | Baseline up to 240 minutes after injection
  Ratio between Standardized uptake values (tumor region) and Standardized uptake values (physiological uptake of brain tissue)
Tumor-to-background ratio on standard scans (60 min after injection) | Baseline up to 60 minutes after injection
  Ratio between Standardized uptake values (tumor region) and Standardized uptake values (physiological uptake of brain tissue)

SECONDARY OUTCOMES:
Standard uptake value comparison | 240 minutes post injection
  Comparison of Standardized uptake values (tumor region) to visual and quantitative parameters on delayed scans (240 min after injection)
Standard uptake value comparison | 60 minutes post injection
  Comparison of Standardized uptake values (tumor region) to visual and quantitative parameters on standard scans (60 min after injection)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States